CLINICAL TRIAL: NCT00354029
Title: Effect of Perioperative i.v. Low-dose S(+) Ketamine in Patients Undergoing Hemorrhoidectomy
Brief Title: Effect of Perioperative i.v. Low-dose S(+) Ketamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Ulrich Johannes Spreng, Asker and Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-001082-41
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Hemorrhoids; Pain
Keywords: hemorrhoids; hemorrhoidectomy; S (+) ketamine; pain
MeSH Terms: conditions — Hemorrhoids; Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Saline 0,9%
  Interventions: Drug: Placebo
- S (+) Ketamine (Active Comparator)
  Interventions: Drug: S (+) Ketamine

INTERVENTIONS:
Drug: S (+) Ketamine — 0,35 mg/kg bolus after induction of anaesthesia; 5 ug/kg/min. continuous until the end of surgery
  Arms: S (+) Ketamine
Drug: Placebo — isotonic saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the use of perioperative intravenous S (+) ketamine reduces the amount and degree of postoperative pain.

Furthermore the purpose of this study is to determine whether the use of perioperative intravenous S (+) ketamine effects cognitive function in the early postoperative period.

DETAILED DESCRIPTION:
The mechanism of development of postoperative pain is complex. Central and peripheral sensitization are playing an important role and this can lead to postoperative hypersensitization. Several studies have shown, that S (+) ketamine can be effective to reduce sensitization and postoperative pain. Ketamine (2-O-chlorophenyl-2-methylamino cyclohexanone) is a N-Methyl-D-Aspartat (NMDA) receptor antagonist. S (+) ketamine has a four times stronger affinity to the NMDA receptor compared to R (-) ketamine. The duration of action for S (+) ketamine is shorter than R (-) ketamine and it has fewer side-effects.

The purpose of this study is to compare the analgetic effect of pregabalin and placebo used in the perioperative period.

The hypothesis is that perioperative intravenous S (+) ketamine gives significant better analgesia than placebo without effecting cognitive function.

The study is including patients undergoing hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of disc prolapse
* Age 18+
* ASA (American Society in Anesthesiology) I-II
* written consent

Exclusion Criteria:

* Age < 18
* ASA > II
* liver failure
* renal failure
* heart failure
* glaucoma
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich J Spreng, Dr. med,, Principal Investigator — Asker and Baerum Hospital, Norway; Vegard Dahl, Dr. med., Study Director — Asker and Baerum Hospital, Norway
Locations (1):
- Asker and Baerum Hospital, Rud, Norway

REFERENCES:
- [Background] Arendt-Nielsen L, Nielsen J, Petersen-Felix S, Schnider TW, Zbinden AM. Effect of racemic mixture and the (S+)-isomer of ketamine on temporal and spatial summation of pain. Br J Anaesth. 1996 Nov;77(5):625-31. doi: 10.1093/bja/77.5.625. PMID 8957979
- [Background] Himmelseher S, Durieux ME. Ketamine for perioperative pain management. Anesthesiology. 2005 Jan;102(1):211-20. doi: 10.1097/00000542-200501000-00030. No abstract available. PMID 15618805
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Peri-operative ketamine for acute post-operative pain: a quantitative and qualitative systematic review (Cochrane review). Acta Anaesthesiol Scand. 2005 Nov;49(10):1405-28. doi: 10.1111/j.1399-6576.2005.00814.x. PMID 16223384

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | S (+) Ketamine | Placebo
Started | 43 | 40
Completed | 39 | 38
Not Completed | 4 | 2
Not completed — Protocol Violation | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S (+) Ketamine | Placebo | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 40 | 83
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.6) | 50.2 (11.4) | 48 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  Norway | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: NRS Pain = Numeric Rating Scale (0-10)
Description: The numeric rating scale (NRS) is used to measure the intensity of pain. The value 0 means no pain and the value 10 represents maximal pain. a higher intensity of pain is associated with a worse outcome.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | S (+) Ketamine | Placebo
Number analyzed (Participants) | 43 | 40
Units on a scale | 1.6 (2.1) | 1.5 (1.7)
Statistical Analysis 1: Comparison: S (+) Ketamine vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | S (+) Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 0/43 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes